CLINICAL TRIAL: NCT03517150
Title: Efficiency of Intraoral Appliance in the Treatment of Obstructive Sleep Apnea Syndrome in Obese Class III
Brief Title: Intraoral Appliance in the Treatment of Obstructive Sleep Apnea Syndrome in Obese
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Silvia de Carvalho Alvarenga, principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FOB apnea
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group will use an oral appliance for treatment of obstructive sleep apnea. The oral appliance is custom-made and its titration is attained by means of progressive mandibular advancement that incrementally moves the mandible forward. This group of patients will use the oral appliance for 45 days.
  Interventions: Device: mandibular advancement device
- Control group (Active Comparator): This group will use a single adjustable silicone appliance in maxillar for 45 days, in order to compare to the experimental group.
  Interventions: Device: mandibular advancement device

INTERVENTIONS:
Device: mandibular advancement device

SUMMARY:
This study evaluates the effectiveness of intraoral appliance in the treatment of obstructive sleep Apnea Syndrome in class III obese in comparison to an adjustable silicone appliance. Both treatments will be test by all of the participants and they will make the polysomnography exam to have the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥40 kg/m² and ≤ 49,9 kg/m²
* Female and male patients (Both of gender patients) with ages between 20 to 65 years old
* Obstructive Sleep Apnea (OSA) diagnosis by polysomnography

Exclusion Criteria:

* sedative drugs users
* Oxygen-dependent or decompensated lung disease
* Decompensated congestive heart failure
* Signs and symptoms of other sleeping disorders (narcolepsy, restless legs syndrome, insomnia)
* craniofacial deformities carriers
* previous OSAS Diagnosis and treatment
* Active Oncological diseases in the last ten years
* Patients with less than 8 teeth per arcade;
* Patients with advanced periodontitis;

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05-12 (Actual); Primary Completion 2018-05-19 (Estimated); Study Completion 2018-06-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 10 minutes
  The Short-Form 36-Item Health Survey (SF-36) will be used to measure quality of life. This instrument will evaluate the physical health component (PHC) and the mental health component (MHC) through the following dimensions: functional capacity, physical aspects, pain, general health status, vitality, social aspects, emotional aspects and mental health.
Daytime sleepiness | 5 minutes
  The Epworth sleepiness scale (ESS) wil measure the subjective daytime sleepiness, assesses the propensity to sleep under inappropriate circumstances. The ESS questionnaire consists of 8 questions about daytime sleepiness in various situations.
Quality of sleep | 5 minutes
  The Pittsburgh Sleep Quality Index is the instrument deployed to evaluate the subjective quality of sleep and the presence of possible disorders. The overall score is formed by the sum of seven components, which can be considered individually, being: 1 - Subjective sleep quality; 2 - sleep latency; 3 - Sleep duration; 4 - Usual efficiency; 5 - Sleep disorders; 6 - Use of sleep medications; 7 - Daytime sleepiness and disturbances during the day. The overall score is formed by the sum of seven components, which can be considered individually, being: 1 - Subjective sleep quality; 2 - sleep latency; 3 - Sleep duration; 4 - Usual efficiency; 5 - Sleep disorders; 6 - Use of sleep medications; 7 - Daytime sleepiness and disturbances during the day. The score is determined by the sum of the seven components, with each answer being given a score between 0 and 3 points. The maximum score of the instrument is 21. The scores> 5 points indicate poor quality in the sleep pattern.

SECONDARY OUTCOMES:
Apnea-hypopnea index (AHI) | 8 hours
  The obstructive Apnea-hypopnea Index is defined as the mean number of obstructive apneas and hypopneas per hour of sleep, thus: the occurrence of 5 to 14 events per hour of sleep means presence of mild apnea, 15 to 29 moderate apnea and ≥ 30 severe apnea. The AHI is derived from overnight polysomnography.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takama N, Kurabayashi M. Influence of untreated sleep-disordered breathing on the long-term prognosis of patients with cardiovascular disease. Am J Cardiol. 2009 Mar 1;103(5):730-4. doi: 10.1016/j.amjcard.2008.10.035. Epub 2009 Jan 12. PMID 19231343
- [Background] Flegal KM, Kit BK, Orpana H, Graubard BI. Association of all-cause mortality with overweight and obesity using standard body mass index categories: a systematic review and meta-analysis. JAMA. 2013 Jan 2;309(1):71-82. doi: 10.1001/jama.2012.113905. PMID 23280227
- [Background] Hamilton GS, Meredith IT, Walker AM, Solin P. Obstructive sleep apnea leads to transient uncoupling of coronary blood flow and myocardial work in humans. Sleep. 2009 Feb;32(2):263-70. doi: 10.1093/sleep/32.2.263. PMID 19238814
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Prospective Studies Collaboration; Whitlock G, Lewington S, Sherliker P, Clarke R, Emberson J, Halsey J, Qizilbash N, Collins R, Peto R. Body-mass index and cause-specific mortality in 900 000 adults: collaborative analyses of 57 prospective studies. Lancet. 2009 Mar 28;373(9669):1083-96. doi: 10.1016/S0140-6736(09)60318-4. Epub 2009 Mar 18. PMID 19299006
- [Background] Tefft BC. Prevalence of motor vehicle crashes involving drowsy drivers, United States, 1999-2008. Accid Anal Prev. 2012 Mar;45:180-6. doi: 10.1016/j.aap.2011.05.028. PMID 22269499
- [Background] Gottlieb DJ, Ellenbogen JM, Bianchi MT, Czeisler CA. Sleep deficiency and motor vehicle crash risk in the general population: a prospective cohort study. BMC Med. 2018 Mar 20;16(1):44. doi: 10.1186/s12916-018-1025-7. PMID 29554902
- [Background] Jurado-Gamez B, Guglielmi O, Gude F, Buela-Casal G. Workplace accidents, absenteeism and productivity in patients with sleep apnea. Arch Bronconeumol. 2015 May;51(5):213-8. doi: 10.1016/j.arbres.2014.07.003. Epub 2014 Aug 13. English, Spanish. PMID 25129165
- [Background] Guglielmi O, Jurado-Gamez B, Gude F, Buela-Casal G. Occupational health of patients with obstructive sleep apnea syndrome: a systematic review. Sleep Breath. 2015 Mar;19(1):35-44. doi: 10.1007/s11325-014-1015-8. Epub 2014 Jun 22. PMID 24952614
- [Background] Watson NF, Badr MS, Belenky G, Bliwise DL, Buxton OM, Buysse D, Dinges DF, Gangwisch J, Grandner MA, Kushida C, Malhotra RK, Martin JL, Patel SR, Quan SF, Tasali E. Recommended Amount of Sleep for a Healthy Adult: A Joint Consensus Statement of the American Academy of Sleep Medicine and Sleep Research Society. Sleep. 2015 Jun 1;38(6):843-4. doi: 10.5665/sleep.4716. PMID 26039963
- [Background] Guglielmi O, Sanchez AI, Jurado-Gamez B, Buela-Casal G, Bardwell WA. [Obesity and sleep quality: the predictors of depression and anxiety in obstructive sleep apnea syndrome patients]. Rev Neurol. 2011 May 1;52(9):515-21. Spanish. PMID 21484722
- [Background] Kern PA, Di Gregorio GB, Lu T, Rassouli N, Ranganathan G. Adiponectin expression from human adipose tissue: relation to obesity, insulin resistance, and tumor necrosis factor-alpha expression. Diabetes. 2003 Jul;52(7):1779-85. doi: 10.2337/diabetes.52.7.1779. PMID 12829646
- [Background] Lee B, Shao J. Adiponectin and energy homeostasis. Rev Endocr Metab Disord. 2014 Jun;15(2):149-56. doi: 10.1007/s11154-013-9283-3. PMID 24170312
- [Background] Ohashi K, Ouchi N, Matsuzawa Y. Anti-inflammatory and anti-atherogenic properties of adiponectin. Biochimie. 2012 Oct;94(10):2137-42. doi: 10.1016/j.biochi.2012.06.008. Epub 2012 Jun 17. PMID 22713764
- [Background] Destors M, Tamisier R, Galerneau LM, Levy P, Pepin JL. [Pathophysiology of obstructive sleep apnea syndrome and its cardiometabolic consequences]. Presse Med. 2017 Apr;46(4):395-403. doi: 10.1016/j.lpm.2016.09.008. Epub 2017 Jan 23. French. PMID 28126503
- [Background] Baron KG, Reid KJ, Kim T, Van Horn L, Attarian H, Wolfe L, Siddique J, Santostasi G, Zee PC. Circadian timing and alignment in healthy adults: associations with BMI, body fat, caloric intake and physical activity. Int J Obes (Lond). 2017 Feb;41(2):203-209. doi: 10.1038/ijo.2016.194. Epub 2016 Oct 31. PMID 27795550
- [Background] Taheri S, Lin L, Austin D, Young T, Mignot E. Short sleep duration is associated with reduced leptin, elevated ghrelin, and increased body mass index. PLoS Med. 2004 Dec;1(3):e62. doi: 10.1371/journal.pmed.0010062. Epub 2004 Dec 7. PMID 15602591
- [Background] Yaggi HK, Araujo AB, McKinlay JB. Sleep duration as a risk factor for the development of type 2 diabetes. Diabetes Care. 2006 Mar;29(3):657-61. doi: 10.2337/diacare.29.03.06.dc05-0879. PMID 16505522
- [Background] Cowan DC, Allardice G, Macfarlane D, Ramsay D, Ambler H, Banham S, Livingston E, Carlin C. Predicting sleep disordered breathing in outpatients with suspected OSA. BMJ Open. 2014 Apr 15;4(4):e004519. doi: 10.1136/bmjopen-2013-004519. PMID 24736037
- [Background] Correa CM, Gismondi RA, Cunha AR, Neves MF, Oigman W. Twenty-four hour Blood Pressure in Obese Patients with Moderate-to-Severe Obstructive Sleep Apnea. Arq Bras Cardiol. 2017 Oct;109(4):313-320. doi: 10.5935/abc.20170130. Epub 2017 Sep 4. PMID 28876375
- [Background] Lopez PP, Stefan B, Schulman CI, Byers PM. Prevalence of sleep apnea in morbidly obese patients who presented for weight loss surgery evaluation: more evidence for routine screening for obstructive sleep apnea before weight loss surgery. Am Surg. 2008 Sep;74(9):834-8. PMID 18807673
- [Background] Bartlett D, Wong K, Richards D, Moy E, Espie CA, Cistulli PA, Grunstein R. Increasing adherence to obstructive sleep apnea treatment with a group social cognitive therapy treatment intervention: a randomized trial. Sleep. 2013 Nov 1;36(11):1647-54. doi: 10.5665/sleep.3118. PMID 24179297
- [Background] Ramar K, Dort LC, Katz SG, Lettieri CJ, Harrod CG, Thomas SM, Chervin RD. Clinical Practice Guideline for the Treatment of Obstructive Sleep Apnea and Snoring with Oral Appliance Therapy: An Update for 2015. J Clin Sleep Med. 2015 Jul 15;11(7):773-827. doi: 10.5664/jcsm.4858. PMID 26094920
- [Background] Battan G, Kumar S, Panwar A, Atam V, Kumar P, Gangwar A, Roy U. Effect of CPAP Therapy in Improving Daytime Sleepiness in Indian Patients with Moderate and Severe OSA. J Clin Diagn Res. 2016 Nov;10(11):OC14-OC16. doi: 10.7860/JCDR/2016/23800.8876. Epub 2016 Nov 1. PMID 28050420
- [Background] Doff MH, Hoekema A, Wijkstra PJ, van der Hoeven JH, Huddleston Slater JJ, de Bont LG, Stegenga B. Oral appliance versus continuous positive airway pressure in obstructive sleep apnea syndrome: a 2-year follow-up. Sleep. 2013 Sep 1;36(9):1289-96. doi: 10.5665/sleep.2948. PMID 23997361
- [Background] Young D, Collop N. Advances in the treatment of obstructive sleep apnea. Curr Treat Options Neurol. 2014 Aug;16(8):305. doi: 10.1007/s11940-014-0305-6. PMID 24957654
- [Background] Wozniak DR, Lasserson TJ, Smith I. Educational, supportive and behavioural interventions to improve usage of continuous positive airway pressure machines in adults with obstructive sleep apnoea. Cochrane Database Syst Rev. 2014 Jan 8;(1):CD007736. doi: 10.1002/14651858.CD007736.pub2. PMID 24399660
- [Background] Dieltjens M, Braem MJ, Vroegop AVMT, Wouters K, Verbraecken JA, De Backer WA, Van de Heyning PH, Vanderveken OM. Objectively measured vs self-reported compliance during oral appliance therapy for sleep-disordered breathing. Chest. 2013 Nov;144(5):1495-1502. doi: 10.1378/chest.13-0613. PMID 23928873
- [Background] Almeida FR, Dal-Fabbro C, Chaves Jr CM. Síndrome da apneia e hipopneia obstrutiva do sono (SAHOS): tratamento com aparelhos intra-orais. In: Tufik, S. Medicina e biologia do sono.1ª ed. São Paulo: Manole; 2008. p. 263-80.
- [Background] Shelgikar AV, Aronovich S, Stanley JJ. Multidisciplinary Alternatives to CPAP Program for CPAP-Intolerant Patients. J Clin Sleep Med. 2017 Mar 15;13(3):505-510. doi: 10.5664/jcsm.6508. PMID 28095977
- [Background] Spicuzza L, Caruso D, Di Maria G. Obstructive sleep apnoea syndrome and its management. Ther Adv Chronic Dis. 2015 Sep;6(5):273-85. doi: 10.1177/2040622315590318. PMID 26336596
- [Background] Chan AS, Sutherland K, Schwab RJ, Zeng B, Petocz P, Lee RW, Darendeliler MA, Cistulli PA. The effect of mandibular advancement on upper airway structure in obstructive sleep apnoea. Thorax. 2010 Aug;65(8):726-32. doi: 10.1136/thx.2009.131094. PMID 20685749
- [Background] Kuhn E, Schwarz EI, Bratton DJ, Rossi VA, Kohler M. Effects of CPAP and Mandibular Advancement Devices on Health-Related Quality of Life in OSA: A Systematic Review and Meta-analysis. Chest. 2017 Apr;151(4):786-794. doi: 10.1016/j.chest.2017.01.020. Epub 2017 Jan 24. PMID 28130044
- [Background] Schwartz M, Acosta L, Hung YL, Padilla M, Enciso R. Effects of CPAP and mandibular advancement device treatment in obstructive sleep apnea patients: a systematic review and meta-analysis. Sleep Breath. 2018 Sep;22(3):555-568. doi: 10.1007/s11325-017-1590-6. Epub 2017 Nov 11. PMID 29129030
- [Background] Sutherland K, Phillips CL, Cistulli PA (2015) Efficacy versus effectiveness in the treatment of obstructive sleep apnea: CPAP and oralappliances.J Dent Sleep Med2:175-181.10.15331/jdsm.5120
- [Background] Haviv Y, Bachar G, Aframian DJ, Almoznino G, Michaeli E, Benoliel R. A 2-year mean follow-up of oral appliance therapy for severe obstructive sleep apnea: a cohort study. Oral Dis. 2015 Apr;21(3):386-92. doi: 10.1111/odi.12291. Epub 2014 Oct 28. PMID 25207802
- [Background] Hoffstein V. Review of oral appliances for treatment of sleep-disordered breathing. Sleep Breath. 2007 Mar;11(1):1-22. doi: 10.1007/s11325-006-0084-8. PMID 17136406
- [Result] AlGhanim N, Comondore VR, Fleetham J, Marra CA, Ayas NT. The economic impact of obstructive sleep apnea. Lung. 2008 Jan-Feb;186(1):7-12. doi: 10.1007/s00408-007-9055-5. Epub 2007 Dec 8. PMID 18066623
- [Result] Anandam A, Akinnusi M, Kufel T, Porhomayon J, El-Solh AA. Effects of dietary weight loss on obstructive sleep apnea: a meta-analysis. Sleep Breath. 2013 Mar;17(1):227-34. doi: 10.1007/s11325-012-0677-3. Epub 2012 Feb 29. PMID 22374151
- [Result] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376
- See also: American Academy of Sleep Medicine — http://www.aasmnet.org/store/product.aspx?pid=10